CLINICAL TRIAL: NCT04851665
Title: Intelligent Cooperation is Influenced by Learning Theories
Status: Withdrawn | Type: Observational
Why Stopped: This was a review of existing de-identified records
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 19-009
Record Dates: First submitted 2021-04-11; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Surgical Education
Keywords: surgical education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention - this was a qualitative analysis — No Intervention - this was a qualitative analysis

SUMMARY:
Qualitative Review of Intraoperative teaching and learning

DETAILED DESCRIPTION:
From manuscript draft Methods:

2.1 Setting, Participants and Data Collection In this qualitative study the investigators examined authentic examples of intraoperative teaching exchanges between attending and resident surgeons. These examples were taken from two previous studies conducted at a large women's hospital: the objectives of those studies were to compare attending and resident responses regarding avoiding intraoperative errors[31] and to develop the previously mentioned Intelligent Cooperation framework.[10] The 10 surgical cases were gynecologic, representing open abdominal, laparoscopic, and vaginal approaches. Surgical cases were chosen by convenience, according to the schedule of the filmographer. Participants included ten surgical attendings, four fellows, and eleven Obstetrics and Gynecology residents, ranging from PGY1 to PGY4. the investigators conducted interviews with all ten attending surgeons and five of the residents. The data for this study included the case video, deidentified transcripts of the cases, and deidentified transcripts of the interviews. Our qualitative approach was most informed by Sandelowski's concept of developing rich qualitative descriptions.[32]

2.2 Research Team the investigators' interdisciplinary research team consisted of a female pelvic surgeon with twenty years of surgical teaching experience (GS), a medical education researcher and educational sociologist (LA), a neurosurgeon and administrator with 30 years of experience across the continuum of medical education (SK), and a cognitive psychologist with expertise in surgical education research (EBL).

2.3 Data Analysis the investigators reviewed and discussed the works of key sociocultural learning scholars, as described in our Introduction. The discussions were converted into a list of "key tenets" of the SCLTs, with associated examples from K-12 and Higher Education. (see Table 1) the investigators then independently coded all transcripts according to the key tenets and examples from our list, noting which exchanges reflected various sociocultural theories. Counting themes was not part of the methodological approach in this study because it was inconsistent with the intent of the study to develop deep, rich, and comprehensive insights about teaching in the OR.[33] the investigators subsequently met as a group to review coding, convert them into themes of teaching and learning advanced surgical skills, and select notable examples from our data. (see Table 2) These themes were then transformed into instructional strategies to improve surgical teaching, based on the sociocultural theories. (see Table 3) Disagreements were settled by group discussion. Data saturation was determined according to our study objective[34], to identify intraoperative instructional strategies related to the social cultural learning theories. the investigators stopped analyzing transcripts when the investigators had generated no new instructional strategies.

2.4 Reflexivity and Ethics During the meetings, the investigators maintained a reflexive atmosphere, reflecting on their backgrounds, experience, and biases and how those might affect their interpretation of the data. the investigators challenged those biases often. the investigators reached consensus regarding differences in data interpretation through group discussion. The University IRB approved this study as exempt.

ELIGIBILITY:
Inclusion Criteria:

Films and transcripts from the database

Exclusion Criteria:

None: the investigators will consider all films and transcripts from the database

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The films included ten surgical attendings, four fellows, and eleven Obstetrics and Gynecology residents, ranging from PGY1 to PGY4. We conducted interviews with all ten attending surgeons and five of the residents.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Themes related to Surgical teaching and learning | approximately 1 year
  Themes were derived by thematic analysis, as informed by Sandelowski's concept of developing rich qualitative descriptions

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT04851665/Prot_000.pdf